CLINICAL TRIAL: NCT05646355
Title: Colorectal Cancer Screening Through Proactive Outreach and Navigation in a Federally Qualified Health Care Center in Brooklyn
Brief Title: Flatbush FHC Proactive Colorectal Cancer Screening and Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-00730
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Screening Outreach (Experimental): Participants will receive a letter from their clinic explaining CRC screening options (fecal immunochemical test (FIT) vs colonoscopy) including a FIT kit with completion and return instructions. The letter will also include information for navigation to a screening colonoscopy instead of FIT testing, if deemed to be the participant's preference.
  Approximately 10-14 days after mailing the FIT kit, participants who have not completed screening will receive a telephone call (with voice message left) and text message, querying whether the FIT kit was received and reminding the participant to complete the test or request a new kit, if needed.
  If the FIT kit has not been submitted after about two weeks from the reminder call/text message, the study team will mail a final letter to the participant on behalf of the clinic, reminding them to complete and return the FIT kit.
  Interventions: Behavioral: Proactive CRC Screening Outreach
- Usual Care (Active Comparator): Individuals in the usual care group will not be approached or notified of their enrollment in the study.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Proactive CRC Screening Outreach — Proactive approach that incorporates a mailed outreach invitation to screen with fecal immunochemical testing (FIT), followed by active assistance to colonoscopy completion if preferred or indicated by FIT test result.
  Arms: Proactive Screening Outreach
Behavioral: Usual Care — Participants will not receive additional outreach from the study team regarding CRC screening.
  Arms: Usual Care

SUMMARY:
The proposed study is a randomized controlled pilot trial designed to assess the effectiveness and acceptability of a proactive screening outreach program on colorectal cancer screening rates on eligible patients in the Flatbush Family Health Center medical practice.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled pilot trial designed to assess the effectiveness and acceptability of a proactive screening outreach program on colorectal cancer screening rates on eligible patients in the Flatbush Family Health Center medical practice, which provides free and subsidized health services to underrepresented minorities. The investigators will randomize patients to the proactive screening outreach arm which will include mailed letters providing patients with information regarding their eligibility for and instructions for performing colorectal cancer screening with FIT testing or colonoscopy. Colorectal cancer screening rates via FIT testing or colonoscopy will be compared in the proactive outreach group and the usual care group. The investigators hypothesize that rates of colorectal cancer screening will improve in underserved populations with the implementation of a proactive approach that incorporates a mailed outreach invitation to screen, followed by active assistance to a colonoscopy completion if preferred or indicated.

ELIGIBILITY:
Inclusion Criteria:

* Receiving medical care at Flatbush FHC
* Due or overdue for CRC screening

Exclusion Criteria:

* Age younger than 45 years old or greater than 75 years old
* Up-to-date with colorectal cancer screening (FIT within 1 year or colonoscopy within 10 years)
* History of colorectal cancer, inflammatory bowel disease or colorectal polyps
* No address or phone number on file
* FIT test ordered within 6 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aasma Shaukat, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Brooklyn Family Health Centers, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Aasma.Shaukat@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Aasma.Shaukat@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Proactive Screening Outreach: Participants will receive a letter from their clinic explaining CRC screening options (fecal immunochemical test (FIT) vs colonoscopy) including a FIT kit with completion and return instructions. The letter will also include information for navigation to a screening colonoscopy instead of FIT testing, if deemed to be the participant's preference.
  Approximately 10-14 days after mailing the FIT kit, participants who have not completed screening will receive a telephone call (with voice message left) and text message, querying whether the FIT kit was received and reminding the participant to complete the test or request a new kit, if needed.
  If the FIT kit has not been submitted after about two weeks from the reminder call/text message, the study team will mail a final letter to the participant on behalf of the clinic, reminding them to complete and return the FIT kit.
  Proactive CRC Screening Outreach: Proactive approach that incorporates a mailed outreach invitation to screen with fecal immunochemical testing (FIT), followed by active assistance to colonoscopy completion if preferred or indicated by FIT test result.
Period: Overall Study
Arm/Group | Proactive Screening Outreach | Usual Care
Started | 59 | 50
Completed | 50 | 50
Not Completed | 9 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — translated materials not available for pilot | 2 | 0
Not completed — no longer screen eligible (completed screening prior to intervention) | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proactive Screening Outreach | Usual Care | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.54 (8.53) | 55.40 (8.42) | 55.47 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 47 | 47 | 94
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 45 | 45 | 90
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Initial Fecal Immunochemical Test (FIT) at 6 Months
Description: Number of Participants who completed CRC screening via FIT by 6 months past the start of intervention
Time Frame: Up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Screening Outreach | Usual Care
Number analyzed (Participants) | 50 | 50
Participants | 7 | 0

2. Primary Outcome: Number of Participants Who Completed Colonoscopy at 6 Months
Description: Number of Participants who underwent colonoscopy by 6 months past the start of intervention
Time Frame: Up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Screening Outreach | Usual Care
Number analyzed (Participants) | 50 | 50
Participants | 4 | 1

3. Secondary Outcome: Number of Participants With Positive FIT Test Who Complete Colonoscopy at 6 Months
Description: Number of Participants who underwent colonoscopy after a positive FIT result by 6 months past the start of intervention
Time Frame: Up to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Screening Outreach | Usual Care
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: This was a pilot offering standard-of-care at-home colorectal cancer screening tests to 50% of the patient population included. No AE or SAE were expected. Although not a study procedure, participants who underwent colonoscopy were systematically assessed for post-procedure events via EMR review, none were observed.
Arm/Group | Proactive Screening Outreach | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT05646355/Prot_SAP_000.pdf